CLINICAL TRIAL: NCT04172753
Title: Feasibility of Imaging and Radiotherapy on a Novel 1.5 T Hybrid Magnetic Resonance Imaging - Linear Accelerator System (MR-Linac)
Brief Title: Feasibility of Online MR-guided Radiotherapy on a 1.5T MR-Linac
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Cihan Gani, Lead of gastrointestinal radiation oncology, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 659/2017BO1
Record Dates: First submitted 2019-11-04; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Rectal Cancer; Head and Neck Cancer; Liver Cancer; Breast Cancer; Prostate Cancer; Oligometastasis; Esophageal Cancer
Keywords: Radiotherapy; Adaptive Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Rectal and anal cancer (Experimental): In this arm patients with rectal and anal cancer are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Prostate cancer (Experimental): In this arm patients with prostate cancer are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Head and neck cancer (Experimental): In this arm patients with head and neck cancers are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Esophageal cancer (Experimental): In this arm patients with esophageal cancer are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Breast Cancer (Experimental): In this arm patients with breast cancer are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Central nervous system tutors (Experimental): In this arm patients with tumors of the central nervous system are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Palliative treatments (Experimental): In this arm patients with palliative treatments are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Other (Experimental): In this arm patients with other tumors are recruited.
  Interventions: Radiation: Radiotherapy on the MR-Linac
- Imaging only (Experimental): In this arm patients receive only imaging on the MR-Linac
  Interventions: Diagnostic Test: Imaging on the MR Linac

INTERVENTIONS:
Radiation: Radiotherapy on the MR-Linac — Radiotherapy is performed on the 1.5 T MR Linac
  Arms: Breast Cancer; Central nervous system tutors; Esophageal cancer; Head and neck cancer; Other; Palliative treatments; Prostate cancer; Rectal and anal cancer
Diagnostic Test: Imaging on the MR Linac — Only imaging performed on the MR Linac
  Arms: Imaging only

SUMMARY:
This study investigates the feasibility of imaging and treatment on a novel 1.5 T MR-Linac radiotherapy hybrid device.

DETAILED DESCRIPTION:
Novel hybrid devices combine magnetic resonance imaging (MRI) and a linear accelerator in a single device. The superior soft tissue contrast compared with cone-beam computed tomography based treatment and the possibility for daily plan adaptation promise a higher precision of treatment, better target volume coverage and normal tissue sparing. In a first step the present study will test the feasibility of imaging and treatment on the 1.5 T MR-Linac.

ELIGIBILITY:
Inclusion Criteria:

* existing indication for radiation therapy
* minimum age 18 years, no upper age limit
* capacity for consent
* Informed consent

Exclusion Criteria:

* contraindication for MRI (claustrophobia, metallic implants not applicable for MRI
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of online MR guided Radiotherapy | During every single patients treatment (i.e. between one to seven weeks after the first application of radiotherapy)
  Treatment of a patient is considered feasible when 85% of treatments were completed as planned in this patient

SECONDARY OUTCOMES:
Time analysis | During every single patients treatment (i.e. between one to seven weeks after the first application of radiotherapy)
  Time required for online MR guided radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Department of Radiation Oncology, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Boeke S, Habrich J, Kubler S, Boldt J, Schick F, Nikolaou K, Kubler J, Gani C, Niyazi M, Zips D, Thorwarth D. Longitudinal assessment of diffusion-weighted imaging during magnetic resonance-guided radiotherapy in head and neck cancer. Radiat Oncol. 2025 Jan 29;20(1):15. doi: 10.1186/s13014-025-02589-9. PMID 39881423
- [Derived] Potkrajcic V, Gani C, Fischer SG, Boeke S, Niyazi M, Thorwarth D, Voigt O, Schneider M, Monnich D, Kubler S, Boldt J, Hoffmann E, Paulsen F, Mueller AC, Wegener D. Online Adaptive MR-Guided Ultrahypofractionated Radiotherapy of Prostate Cancer on a 1.5 T MR-Linac: Clinical Experience and Prospective Evaluation. Curr Oncol. 2024 May 9;31(5):2679-2688. doi: 10.3390/curroncol31050203. PMID 38785484